CLINICAL TRIAL: NCT05145296
Title: Non-Randomized, Single-Center Pilot Trial Assessing The Safety/Efficacy Of Targeting Peripheral And Central Humoral Alloimmune Memory With Daratumumab And With Belatacept In Highly HLA-Sensitized Patients Awaiting Kidney Transplantation
Brief Title: The Safety/Efficacy Of Daratumumab With Belatacept In Highly HLA-Sensitized Patients Awaiting Kidney Transplantation
Acronym: COMBAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: limited clinically significant reduction on global cPRA levels (access to transplantation was unchanged), as well as restrictions in belatacept supply.
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC21.171
Record Dates: First submitted 2021-10-21; First posted 2021-12-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2023-05

CONDITIONS: Sensitisation; Highly Sensitised Dialysis Patients
Keywords: Highly sensitized kidney transplant; Desensitization; BELATACEPT; Daratumumab
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with cPRA ≥99% (Other): This is a non-randomized, single arm study, combination trial designed according to the Recommendations of the Clinical Trial Design Task Force of the NCI Investigational Drug Steering Committee. The study will enroll 12 patients with cPRA ≥99% on the deceased donor kidney transplant waiting list, who have not received a compatible donor offer for >3 year. According to inclusion and exclusion criteria patients will be screened to participate in the trial.
  Interventions: Combination Product: Each patient will undergo in the first step of the study belatacept treatment and in the second apheresis and daratumumab

INTERVENTIONS:
Combination Product: Each patient will undergo in the first step of the study belatacept treatment and in the second apheresis and daratumumab — Four consecutive cohorts each comprising 3 patients are planned. STEP I: Patients receive Belatacept 10mg/kg, administered on days 1, 5, end of week 2, 4 and 8 .
  Patients without a significant decrease in the global cPRA (cPRA or TGI ≥99%) or significant reduction of anti-HLA Ab MF will continue to the second step.
  STEP II: (15 weeks) One week after the last injection of belatacept, patients will undergo 4 sessions of apheresis (plasmapheresis (PF) or Immunoadsorption (IA)) which will be given every 48h. At week 11, patients will receive 4 doses of daratumumab (8mg/kg) every two weeks until week 17. Daratumumab will be alternated with 4 additional doses of belatacept 5 mg/kg FOLLOW-UP (24 weeks) All patients exiting the study, either having completed all treatment courses or exiting prematurely (transplanted or not), will be proposed monthly follow-up visits
  Other Names: combination trial designed

SUMMARY:
While the number of kidney transplants is increasing worldwide every year, there is a clear imbalance between the high number of patients in the waiting list and those receiving a transplant and importantly, among waitlist patients there is a progressively higher number of highly sensitised patients that have very low or even no chance to receive a compatible organ. These patients remain for very long periods of time on dialysis therapy, having lower quality of life, lower life expectancy and produce higher health-related costs. Unfortunately, current desensitization therapies have shown very poor success and patients usually lose these grafts very fast if transplanted across a positive cross-match. Therefore, there is an urgent need for novel desensitization strategies capable of overcoming this immunological barrier and allow an increasing number of patients to receive a HLA-compatible kidney allograft.This is a non-randomized, single arm study, combination trial designed according to the Recommendations of the Clinical Trial Design Task Force of the NCI Investigational Drug Steering Committee. The study will enroll 12 patients with cPRA or TGI ≥99% on the deceased donor kidney transplant waiting list, who have not received a compatible donor offer for >3 year. According to inclusion and exclusion criteria patients will be screened to participate in the trial.

DETAILED DESCRIPTION:
This is a non-randomized, single arm study, combination trial designed according to the Recommendations of the Clinical Trial Design Task Force of the NCI Investigational Drug Steering Committee. The study will enroll 12 patients with cPRA or TGI ≥99% on the deceased donor kidney transplant waiting list, who have not received a compatible donor offer for >3 year. According to inclusion and exclusion criteria patients will be screened to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-70 years
* End Stage Renal Disease (ESRD) on dialysis
* Patient listed and active for a deceased donor kidney transplant and have not received compatible donor offer for ≥3 year.
* Calculated PRA ≥ 99%
* Positive CMV serology
* Positive EBV serology
* Current vaccination for more than one month for diphtheria, tetanus, poliomyelitis, influenza, pneumococcus, meningococcus, herpes zoster and SARS CoV-2.
* Patient affiliated to social security insurance or beneficiary of social security insurance

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol

  * Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including HIV, hepatitis B, hepatitis C, zoster)
  * Patient with positive hepatitis core antigen and/or positive hepatitis B surface antigen
  * Serious uncontrolled concomitant major organ disease
  * Any infection requiring hospitalization and intravenous antibiotics within 4 weeks of screening or Per os antibiotics within 2 weeks
  * Primary or secondary immunodeficiency
  * History of active tuberculosis (TB) (even if treated) or untreated latent TB
  * Malignancy within the last 5 years except documented and treated basal and squamous cell cancer of the skin
  * Alcohol, drug or chemical abuse within 1 year
  * Difficult peripheral venous access
  * Negative EBV serology
  * Negative CMV serology
  * Neutropenia (ANC <1000/uL) or thrombocytopenia (platelet count <100,000/uL) within 4 weeks prior to study entry
  * Patient previously treated with investigational products (belatacept, daratumumab)
  * Severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
  * Hypersensitivity to any active substance or component of the investigational medicinal products
  * Any contra-indication to premedication drugs (paracetamol, dexchlorpheniramine, cetirizine, dexamethasone, montelukast) or post-medication drugs (corticosteroids, bronchodilators, valaciclovir)
  * Immunization with live vaccine within 2 months of study entry
  * Dry body weight ≥75kg.
  * Pregnancy or lactation
  * Females with childbearing status, defined as a premenopausal female capable of becoming pregnant, and not using an effective form of birth control. Effective birth control methods include oral, implant or patch hormone contraception; intrauterine device; abstinence and outercourse; tubal ligation; vasectomy.
  * Participant involved in another interventional clinical study
  * Person deprived of liberty by judicial order
  * Person under guardianship or curatorship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Proportion of severe or medically significant Adverse and Serious Adverse Events | end of study
  Proportion of severe or medically significant Adverse and Serious Adverse Events, defined by:
  Any grade 3 or higher infection (according to the CTCAE definition, i.e. IV antibiotic, antifungal, or antiviral intervention indicated; or invasive intervention indicated) during the interventional study period (6 months).
  Success will be defined by a proportion of toxicity below 17% (≤2/12).

SECONDARY OUTCOMES:
Assess the efficacy of dual targeting with anti-CD38 mAb daratumumab (Darzalex®) and co-stimulation blockade with belatacept (Nulojix®) in HLA-sensitized patients | end of study
  Proportion of patients in whom ≥10 HLA antibodies (class I and/or class II) are eliminated (undetectable or <2000 MFI) OR cPRA(or TGI) decrease to <99% at the end of step I and at the end of step II.
  Success will be defined by an efficacy of 66% (≥8/12)
Evaluate the impact of belatacept on anti-HLA antibody reduction using single antigen beads (SAB) in terms of MFI and specificities | Week 9
  Total number and mean number of HLA antibodies at the end of Step I (belatacept) as compared to baseline
Evaluate the impact of belatacept on circulating Tfh cells compared to baseline belatacept therapy and at the end of this therapy (Step I). | week 9 compared to baseline
  Change in number and percentages of subtypes of circulating Peripheral T helper cells (TPH) including Tfh cells at the end of belatacept therapy
Evaluate the impact of belatacept on circulating HLA-specific mBC and their capacity to produce anti-HLA antibodies as well as numbers function of HLA-specific LLPC in bone marrow compared to baseline therapy and at the end of this therapy (Step I) | Week 9
  Proportion of patients with a reduction of circulating HLA-specific memory B cells (both class I and class II)
Evaluate the impact of the dual combination of belatacept and daratumumab on anti-HLA antibody reduction using single antigen beads (SAB) in terms of MFI and specificities | week 24 compared to baseline
  Change in number and mean number of HLA antibodies at the end of Step II (belatacept followed by daratumumab)
Evaluate the impact of the dual combination of belatacept and daratumumab on circulating Tfh cells compared to baseline and the end of this dual therapy and at the time of a kidney transplantation, if any (Step II). | week 24 compared to baseline
  Change in number and percentages of subtypes of circulating Tfh cells at the end of dual therapy and at the time of an kidney transplantation as compared to baseline
Evaluate the impact of the dual combination of belatacept and daratumumab on circulating HLA-specific mBc and their capacity to produce anti-HLA antibodies as well as numbers and function of LLPC in bone marrow compared to baseline and the end of this | week 24
  Proportion of patients with a reduction of circulating HLA-specific memory B cells (both class I and class II)
Evaluate the impact of the dual combination of belatacept and daratumumab on immunodominant HLA antibody (class I and Class II) at the end Step II as compared to baseline and as compared to the end of Step I | week 24
  Mean reduction in MFI of the immunodominant HLA antibody, class I and Class II at the end Step II
Evaluate the impact of the dual combination of belatacept and daratumumab on HLA-specific Antibody secreting cells (ASC) frequencies in bone marrow aspirates at the end of Step II as compared to baseline | week 24
  Proportion of patients with a reduction of HLA-specific ASC frequencies in bone marrow aspirates
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | End of study
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0'
Evaluate the impact of the dual combination of belatacept and daratumumab on patients transplanted with a compatible donor | week 18, week 24
  Proportion of patients transplanted with a compatible donor
In case of kidney transplantation, investigate the germinal center activation of iliac lymph nodes obtained at the time of kidney transplantation | day of transplantation
  At the time of kidney transplantation investigate the germinal center activation of iliac lymph nodes obtained during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Malvezzi, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble, La Tronche, France

REFERENCES:
- [Background] Loupy A, Lefaucheur C. Antibody-Mediated Rejection of Solid-Organ Allografts. N Engl J Med. 2018 Sep 20;379(12):1150-1160. doi: 10.1056/NEJMra1802677. No abstract available. PMID 30231232
- [Background] Pruthi R, Hilton R, Pankhurst L, Mamode N, Hudson A, Roderick P, Ravanan R. UK Renal Registry 16th annual report: chapter 4 demography of patients waitlisted for renal transplantation in the UK: national and centre-specific analyses. Nephron Clin Pract. 2013;125(1-4):81-98. doi: 10.1159/000360023. Epub 2014 Feb 14. PMID 24662168
- [Background] Wiebe C, Tambur A, Nickerson PW. A call to action-The transplant recipient's expectation of precision in transplant medicine. Am J Transplant. 2018 Dec;18(12):2845-2846. doi: 10.1111/ajt.15027. Epub 2018 Aug 13. No abstract available. PMID 30022602
- [Background] Kiernan JJ, Ellison CA, Tinckam KJ. Measuring alloantibodies: a matter of quantity and quality. Curr Opin Organ Transplant. 2019 Feb;24(1):20-30. doi: 10.1097/MOT.0000000000000593. PMID 30507703
- [Background] Djamali A, Kaufman DB, Ellis TM, Zhong W, Matas A, Samaniego M. Diagnosis and management of antibody-mediated rejection: current status and novel approaches. Am J Transplant. 2014 Feb;14(2):255-71. doi: 10.1111/ajt.12589. Epub 2014 Jan 8. PMID 24401076
- [Background] Formica RN Jr, Kulkarni S. Being Thoughtful about Desensitization. Clin J Am Soc Nephrol. 2017 Nov 7;12(11):1878-1880. doi: 10.2215/CJN.09000817. Epub 2017 Oct 3. No abstract available. PMID 28974523
- [Background] Cornell LD, Schinstock CA, Gandhi MJ, Kremers WK, Stegall MD. Positive crossmatch kidney transplant recipients treated with eculizumab: outcomes beyond 1 year. Am J Transplant. 2015 May;15(5):1293-302. doi: 10.1111/ajt.13168. Epub 2015 Mar 2. PMID 25731800
- [Background] Luque S, Lucia M, Crespo E, Jarque M, Grinyo JM, Bestard O. A multicolour HLA-specific B-cell FluoroSpot assay to functionally track circulating HLA-specific memory B cells. J Immunol Methods. 2018 Nov;462:23-33. doi: 10.1016/j.jim.2018.07.011. Epub 2018 Jul 31. PMID 30075182
- [Background] Lucia M, Luque S, Crespo E, Melilli E, Cruzado JM, Martorell J, Jarque M, Gil-Vernet S, Manonelles A, Grinyo JM, Bestard O. Preformed circulating HLA-specific memory B cells predict high risk of humoral rejection in kidney transplantation. Kidney Int. 2015 Oct;88(4):874-87. doi: 10.1038/ki.2015.205. Epub 2015 Jul 15. PMID 26176829
- [Background] Perry DK, Pollinger HS, Burns JM, Rea D, Ramos E, Platt JL, Gloor JM, Stegall MD. Two novel assays of alloantibody-secreting cells demonstrating resistance to desensitization with IVIG and rATG. Am J Transplant. 2008 Jan;8(1):133-43. doi: 10.1111/j.1600-6143.2007.02039.x. PMID 18184311
- [Background] Moreno Gonzales MA, Gandhi MJ, Schinstock CA, Moore NA, Smith BH, Braaten NY, Stegall MD. 32 Doses of Bortezomib for Desensitization Is Not Well Tolerated and Is Associated With Only Modest Reductions in Anti-HLA Antibody. Transplantation. 2017 Jun;101(6):1222-1227. doi: 10.1097/TP.0000000000001330. PMID 27379560
- [Background] Kwun J, Burghuber C, Manook M, Iwakoshi N, Gibby A, Hong JJ, Knechtle S. Humoral Compensation after Bortezomib Treatment of Allosensitized Recipients. J Am Soc Nephrol. 2017 Jul;28(7):1991-1996. doi: 10.1681/ASN.2016070727. Epub 2017 Feb 23. PMID 28232617
- [Background] Chen J, Yin H, Xu J, Wang Q, Edelblum KL, Sciammas R, Chong AS. Reversing endogenous alloreactive B cell GC responses with anti-CD154 or CTLA-4Ig. Am J Transplant. 2013 Sep;13(9):2280-92. doi: 10.1111/ajt.12350. Epub 2013 Jul 15. PMID 23855587
- [Background] Yang J, Chen J, Young JS, Wang Q, Yin D, Sciammas R, Chong AS. Tracing Donor-MHC Class II Reactive B cells in Mouse Cardiac Transplantation: Delayed CTLA4-Ig Treatment Prevents Memory Alloreactive B-Cell Generation. Transplantation. 2016 Aug;100(8):1683-91. doi: 10.1097/TP.0000000000001253. PMID 27362308
- [Background] Kim EJ, Kwun J, Gibby AC, Hong JJ, Farris AB 3rd, Iwakoshi NN, Villinger F, Kirk AD, Knechtle SJ. Costimulation blockade alters germinal center responses and prevents antibody-mediated rejection. Am J Transplant. 2014 Jan;14(1):59-69. doi: 10.1111/ajt.12526. PMID 24354871
- [Background] Leibler C, Thiolat A, Henique C, Samson C, Pilon C, Tamagne M, Pirenne F, Vingert B, Cohen JL, Grimbert P. Control of Humoral Response in Renal Transplantation by Belatacept Depends on a Direct Effect on B Cells and Impaired T Follicular Helper-B Cell Crosstalk. J Am Soc Nephrol. 2018 Mar;29(3):1049-1062. doi: 10.1681/ASN.2017060679. Epub 2018 Jan 10. PMID 29321143
- [Background] Leibler C, Matignon M, Pilon C, Montespan F, Bigot J, Lang P, Carosella ED, Cohen J, Rouas-Freiss N, Grimbert P, Menier C. Kidney transplant recipients treated with belatacept exhibit increased naive and transitional B cells. Am J Transplant. 2014 May;14(5):1173-82. doi: 10.1111/ajt.12721. Epub 2014 Apr 14. PMID 24730563
- [Background] Vincenti F, Rostaing L, Grinyo J, Rice K, Steinberg S, Gaite L, Moal MC, Mondragon-Ramirez GA, Kothari J, Polinsky MS, Meier-Kriesche HU, Munier S, Larsen CP. Belatacept and Long-Term Outcomes in Kidney Transplantation. N Engl J Med. 2016 Jan 28;374(4):333-43. doi: 10.1056/NEJMoa1506027. PMID 26816011
- [Background] Bray RA, Gebel HM, Townsend R, Roberts ME, Polinsky M, Yang L, Meier-Kriesche HU, Larsen CP. Posttransplant reduction in preexisting donor-specific antibody levels after belatacept- versus cyclosporine-based immunosuppression: Post hoc analyses of BENEFIT and BENEFIT-EXT. Am J Transplant. 2018 Jul;18(7):1774-1782. doi: 10.1111/ajt.14738. Epub 2018 Apr 17. PMID 29573335
- [Background] Kwun J, Burghuber C, Manook M, Ezekian B, Park J, Yoon J, Yi JS, Iwakoshi N, Gibby A, Hong JJ, Farris AB, Kirk AD, Knechtle SJ. Successful desensitization with proteasome inhibition and costimulation blockade in sensitized nonhuman primates. Blood Adv. 2017 Oct 26;1(24):2115-2119. doi: 10.1182/bloodadvances.2017010991. eCollection 2017 Nov 14. PMID 29296858
- [Background] Alishetti S, Farr M, Jennings D, Serban G, Uriel N, Sayer G, Vasilescu R, Restaino S, Chong AS, Habal MV. Desensitizing highly sensitized heart transplant candidates with the combination of belatacept and proteasome inhibition. Am J Transplant. 2020 Dec;20(12):3620-3630. doi: 10.1111/ajt.16113. Epub 2020 Jul 7. PMID 32506824
- [Background] Jain D, Rajab A, Young JS, Yin D, Nadasdy T, Chong AS, Pelletier RP. Reversing donor-specific antibody responses and antibody-mediated rejection with bortezomib and belatacept in mice and kidney transplant recipients. Am J Transplant. 2020 Oct;20(10):2675-2685. doi: 10.1111/ajt.15881. Epub 2020 Apr 28. PMID 32243663
- [Background] Moreno L, Perez C, Zabaleta A, Manrique I, Alignani D, Ajona D, Blanco L, Lasa M, Maiso P, Rodriguez I, Garate S, Jelinek T, Segura V, Moreno C, Merino J, Rodriguez-Otero P, Panizo C, Prosper F, San-Miguel JF, Paiva B. The Mechanism of Action of the Anti-CD38 Monoclonal Antibody Isatuximab in Multiple Myeloma. Clin Cancer Res. 2019 May 15;25(10):3176-3187. doi: 10.1158/1078-0432.CCR-18-1597. Epub 2019 Jan 28. PMID 30692097
- [Background] Kwun J, Matignon M, Manook M, Guendouz S, Audard V, Kheav D, Poullot E, Gautreau C, Ezekian B, Bodez D, Damy T, Faivre L, Menouche D, Yoon J, Park J, Belhadj K, Chen D, Bilewski AM, Yi JS, Collins B, Stegall M, Farris AB, Knechtle S, Grimbert P. Daratumumab in Sensitized Kidney Transplantation: Potentials and Limitations of Experimental and Clinical Use. J Am Soc Nephrol. 2019 Jul;30(7):1206-1219. doi: 10.1681/ASN.2018121254. Epub 2019 Jun 21. PMID 31227636
- [Background] Paller CJ, Bradbury PA, Ivy SP, Seymour L, LoRusso PM, Baker L, Rubinstein L, Huang E, Collyar D, Groshen S, Reeves S, Ellis LM, Sargent DJ, Rosner GL, LeBlanc ML, Ratain MJ. Design of phase I combination trials: recommendations of the Clinical Trial Design Task Force of the NCI Investigational Drug Steering Committee. Clin Cancer Res. 2014 Aug 15;20(16):4210-7. doi: 10.1158/1078-0432.CCR-14-0521. PMID 25125258
- See also: EMA Summary of product characteristics - Nulojix. — https://www.ema.europa.eu/en/documents/product-information/nulojix-epar-product-information_en.pdf
- See also: EMA Summary of product characteristics - Darzalex. — http://www.ema.europa.eu/en/documents/product-information/darzalex-epar-product-information_en.pdf
- See also: 1. Global Observatory on Donation and Transplantation. GODT at <http://www.transplant-observatory.org/> — https://clinicaltrials.gov/ct2/show/NCT04204980
- See also: Global Observatory on Donation and Transplantation. GODT — http://www.transplant-observatory.org/